CLINICAL TRIAL: NCT03640598
Title: Ultrasound Guided Erector Spinae Versus Ilioinguinal/ Ilio-hypogastric Block for Postoperative Analgesia in Children Undergoing Inguinal Surgeries
Brief Title: Erector Spinae Versus Ilioinguinal/ Ilio-hypogastric Block in Children Undergoing Inguinal Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: R.18.05.202
Record Dates: First submitted 2018-08-18; First posted 2018-08-21 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ilioinguinal/iliohypogastric nerve blocks (Other): The patient will receive ultrasound-guided Ilioinguinal/iliohypogastric nerve blocks
  Interventions: Procedure: Ilioinguinal/iliohypogastric nerve blocks
- Erector spinae nerve block (Other): The patient will receive ultrasound-guided erector spinae nerve block
  Interventions: Procedure: Erector spinae nerve block

INTERVENTIONS:
Procedure: Ilioinguinal/iliohypogastric nerve blocks — The patient will receive ultrasound-guided Ilioinguinal/iliohypogastric nerve blocks with0.5 ml/kg 0.125 mg/kg bupivacaine + fentanyl 2ug/ml injectate
  Arms: Ilioinguinal/iliohypogastric nerve blocks
Procedure: Erector spinae nerve block — The patient will receive ultrasound-guided erector spinae nerve block 0.5 ml/kg 0.125 bupivacaine + fentanyl 2ug/ml injectate.
  Arms: Erector spinae nerve block

SUMMARY:
Investigators aim to compare the efﬁcacy of US-guided II/IH nerve block versus US-guided ES block for pediatric unilateral inguinal hernia repair with respect to postoperative analgesia

DETAILED DESCRIPTION:
regarding patient registry; a prior G power analysis was done. 24 per group was determined to achieve 80% power to detect a difference of 60 min in time to first rescue analgesia between the two groups with a significance level (α) of 0.05 using a two-sided two-sample t-test; 25 patients were included per group to replace any dropouts.

- Statistical analysis: Data will be analyzed through SPSS (Statistical Package for Social Sciences). Program version 22. Distribution of data will be first tested by the Shapiro test. Data will be presented as the mean and standard deviation (SD), median and range or numbers and percentages. For normally distributed data, the unpaired t-test will be used to compare the mean values of both groups. For pain score, Mann Whitney U test will be used. Fisher's exact test will be used for comparison of categorical data. The P value ≤ 0.05 will be considered as the level of statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* : American Society of Anesthesiologists physical status I - II

Exclusion Criteria:

* History of clinically significant cardiac disease.
* History of clinically significant hepatic disease.
* History of clinically significant renal disease.
* History of clinically significant neurological disease.
* Known allergy to local anaesthetics

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2018-10-20 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Postoperative CHEOPS scale | for 6 hours after surgery
  The scale includes six entries with an appropriate point evaluation focused on the character of crying (1-3 points), facial expressions (0-2 points), verbal reaction (0-2 points), position of the body (1-2 points), touch (1-2 points), and position of the legs (1-2 points). Minimum score is 4 (no pain) and maximum is 13 (maximum pain). Grades are summed together. CHEOPS has a minimum possible score of 4 points (no pain) to a maximum of 13 points (the worst pain).
  When the postoperative pain score exceeded four, rescue analgesia was given with a 20mg/kg paracetamol suppository.

SECONDARY OUTCOMES:
Time to first analgesic request | during first 24 hours
  Time to first analgesic request
number of patients requiring rescue analgesic | during first 24 hours
incidence of postoperative nausea and vomiting | during first 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Enas A Abd el Motlb, MD, Study Chair — Assistant Professor, Anesthesia Department
Locations (1):
- Enas A Abd el Motlb, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Undecided